CLINICAL TRIAL: NCT00672867
Title: A Open Randomized Clinical Trial Comparing the Efficacy and Safety of Clevudine 30mg Versus Adefovir 10mg in Patients With LC-B
Brief Title: A Pilot Study to Evaluate the Safety and Efficacy of Clevudine or Adefovir Patients With LC-B
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Bukwang Pharmaceutical (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: L-FMAU-309
Record Dates: First submitted 2008-05-02; First posted 2008-05-06 (Estimated); Last update posted 2014-12-18 (Estimated); Status verified 2012-07

CONDITIONS: Patients With LC-B
MeSH Terms: interventions — clevudine; adefovir dipivoxil

ARMS (2):
- 1 (Experimental): Clevudine
  Interventions: Drug: Clevudine
- 2 (Active Comparator): Adefovir
  Interventions: Drug: Adefovir dipivoxil

INTERVENTIONS:
Drug: Clevudine — 30mg
  Other Names: Levovir
  Arms: 1
Drug: Adefovir dipivoxil — 10mg
  Other Names: Hepsera
  Arms: 2

SUMMARY:
The purpose of this study is to compare the safety and antiviral activity of Clevudine Versus Adefovir dipivoxil in patients with LC-B.

ELIGIBILITY:
Inclusion Criteria:

1. Patient is 18 years and older.
2. 5 ≦ Child-Pugh score ≦ 12
3. Patient is HBV DNA positive with DNA levels ≥ 1 x 10(4) copies/mL within 30 days of baseline.
4. Patient is documented to be HBsAg positive for > 6 months.
5. Patient is HBeAg positive or negative.
6. Patient has ALT or AST levels which are in the range of > 1 x ULN and < 15 X ULN
7. Patient with liver cirrhosis diagnosed by imaging study within 1 year or clinical evidence of portal hypertension
8. Life expectancy of at least 12 months
9. Female patient with a negative urine(Beta-HCG) pregnancy test taken within 14 days of starting therapy.
10. Patient who is able to give written informed consent prior to study start and to comply with the study requirements.

Exclusion Criteria:

1. Patient is currently receiving antiviral, immunomodulatory, cytotoxic or corticosteroid therapy.
2. Previous treatment with interferon must have ended at least 6 months prior to the screening visit.
3. Patients previously treated with clevudine, entecavir, lamivudine, adefovir, telbivudine or any other investigational nucleoside for HBV infection.
4. Patient is coinfected with HCV, HDV or HIV.
5. Patient with clinical evidence of hepatocellular carcinoma
6. Patient has alpha-fetoprotein > 400ng/mL.
7. Patient has Hemoglobin <8g/dL (Male), 7.5g/dL (Female) or WBC <1,500mm3 or Neutrophils <500/mm3 or Platelet count <30,000/mm3.
8. Patient is pregnant or breast-feeding.
9. Patient is unwilling to use an "effective" method of contraception during the study and for up to 3 months after the use of study drug ceases.
10. Patient has a clinically relevant history of abuse of alcohol or drugs.
11. Patient with previous liver transplantation
12. Patient has a significant immunocompromised, gastrointestinal, renal, hematological, psychiatric, bronchopulmonary, biliary diseases excluding asymptomatic GB stone, neurological, cardiac, oncologic(except HCC)or allergic disease or medical illness that in the investigator's opinion might interfere with therapy.
13. Patient has creatinine clearance less than 60mL/min as estimated by the following formula: (140-age in years) (body weight [kg])/(72) (serum creatinine [mg/dL]) [Note: multiply estimates by 0.85 for women]

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 102 (Estimated)
Dates: Start 2007-12; Primary Completion 2012-11 (Actual); Study Completion 2014-09 (Actual)

PRIMARY OUTCOMES:
Proportion of patients with HBV DNA below 12 IU/mL by Real-Time PCR

SECONDARY OUTCOMES:
The change of HBV DNA from the baseline.
Child-Pugh score improvement
MELD score improvement
Biochemical improvement
Proportion of patients with HBeAg loss and/or seroconversion

CONTACTS AND LOCATIONS:
Locations (1):
- Samsung Medical Center, Seoul, South Korea